CLINICAL TRIAL: NCT04614025
Title: A Randomized, Controlled, Multicenter, Parallel-Group Phase IIa Study to Evaluate the Efficacy and Safety of Intramuscular Injections of PLX-PAD for the Treatment of Severe COVID-19
Brief Title: Open-label Multicenter Study to Evaluate the Efficacy of PLX-PAD for the Treatment of COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The decision to bring the Study to early clinical readout came in response to COVID-19's evolution as a disease, and the significant changes in the standard of care, leading to an increase in the severity of conditions of the intubated patients.
Sponsor: Pluristem Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLX-COV-03
Record Dates: First submitted 2020-11-02; First posted 2020-11-03 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: COVID; ARDS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PLX-PAD Treatment (Experimental): PLX-PAD 300 million cells (20 million/mL) administered via 15 IM injections (1 mL each).
  Single administration in addition to best standard medical care.
  Interventions: Biological: PLX-PAD
- Control Group (No Intervention): Best standard medical care

INTERVENTIONS:
Biological: PLX-PAD — PLX-PAD - allogeneic ex-vivo expanded placental mesenchymal-like adherent stromal cells
  Arms: PLX-PAD Treatment

SUMMARY:
This clinical trial will examine if a new treatment of Mesenchymal-like Adherent stromal Cells (called PLX-PAD) can help patients intubated and mechanically ventilated due to COVID-19 to recover more quickly with less complications.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent, or with a legal representative who can provide informed consent.
* Male or non-pregnant female adult 18-85 years of age at time of enrollment.
* Laboratory-confirmed SARS-CoV-2 infection as determined by PCR, in any specimen up to 21 days prior to randomization.
* Meets definition of ARDS according to Berlin criteria.

Key Exclusion Criteria:

* Body weight under 55 kg (121 lbs)
* Serum creatinine level of over 1.5 mg/dL at time of randomization.
* Total Bilirubin ≥2 mg/dL at time of randomization.
* Known allergy to any of the following: dimethyl sulfoxide (DMSO), human serum albumin, bovine serum albumin.
* Stroke or acute myocardial infarction/unstable angina within 3 months prior to randomization.
* Chronic Obstructive Pulmonary disease GOLD stage above II.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Number of ventilator-free days | 28 days

SECONDARY OUTCOMES:
All-cause mortality | 28 and 60 days
Duration of mechanical ventilation | 28 and 60 days

CONTACTS AND LOCATIONS:
Locations (9):
- Germany (4):
  - Charite Campus Virchow, Berlin
  - Campus Benjamin Franklin - CBF Charité - Universitätsmedizin, Berlin
  - University of hospital Bonn, Bonn
  - Hospital Cologne-Merheim, Cologne
- Israel (5):
  - Emek Medical Center, Afula
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Galilee Medical Center, Nahariya
  - Baruch Padeh Medical Center, Poriya, Tiberias

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.pluristem.com